CLINICAL TRIAL: NCT00901693
Title: An Evaluation of the Efficacy and Safety of AL-46383A Ophthalmic Solution for the Treatment of Adenoviral Conjunctivitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Internal business decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-07-53
Record Dates: First submitted 2009-05-08; First posted 2009-05-14 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Adenoviral Conjunctivitis
Keywords: pink eye; eye infection; conjunctivitis
MeSH Terms: conditions — Conjunctivitis; Eye Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AL-46383A (Experimental): AL-46383A Ophthalmic Solution, 1 drop in each eye, 8 times a day for 10 days
  Interventions: Drug: AL-46383A Ophthalmic Solution
- Vehicle (Placebo Comparator): AL-46383A Ophthalmic Solution Vehicle, 1 drop in each eye, 8 times a day, for 10 days
  Interventions: Drug: AL-46383A Ophthalmic Solution Vehicle

INTERVENTIONS:
Drug: AL-46383A Ophthalmic Solution
  Arms: AL-46383A
Drug: AL-46383A Ophthalmic Solution Vehicle
  Arms: Vehicle

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of AL-46383A Ophthalmic Solution for the treatment of adenoviral conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* At least one eye must have EITHER a positive adenovirus test (using the Adeno Detector™ for Adenoviral Conjunctivitis, Rapid Pathogen Screening, Inc.) OR a positive clinical diagnosis assessed by the Adenoviral Clinical Diagnostic Checklist.
* Onset and development of ocular symptoms and/or signs of conjunctivitis ≤ 7 days prior to enrollment (Day 1) in either eye.
* Able to understand and sign an informed consent form that has been approved by an Institutional Review Board/ Independent Ethics Committee (IRB/IEC).
* Must agree to comply with the visit schedule and other requirements of the study.
* Females who are not pregnant and are not lactating. All females of childbearing potential (those who are not pre-menarcheal, not postmenopausal or surgically sterile) may participate only if they have a negative urine pregnancy test prior to randomization, and if they agree to use adequate birth control methods to prevent pregnancy throughout the study.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Sub-epithelial infiltrates at the Day 1 visit in either eye.
* Corneal opacity or any corneal abnormality at the Day 1 visit in either eye.
* Contact lens wear during the course of the study. Participants requiring correction must have spectacles with appropriate correction.
* Only one sighted eye or vision in either eye not correctable to 0.6 or better logMAR (using ETDRS chart) at the Day 1 visit.
* Abnormal findings in the posterior pole of the retina or any media opacity found in a dilated fundus examination at the Day 1 (Screening/ Baseline) visit.
* Suspected fungal, herpes, Chlamydia or Acanthamoeba infection, based on clinical observation.
* History of active uveitis or iritis in either eye.
* History of corneal transplant in either eye.
* Presence of nasolacrimal duct obstruction at Day 1.
* Use of specified prohibited medications.
* Other protocol-defined exclusion criteria may apply.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Sustained microbiological success at Day 5 or Day 7 | Up to Day 18

SECONDARY OUTCOMES:
Time to sustained microbiological success | Up to Day 18

CONTACTS AND LOCATIONS:
Overall Officials: Sally Scheib, Study Director — Alcon Research